CLINICAL TRIAL: NCT06337344
Title: Enhanced Executive Functioning After Single-session Mind-body Practice is Associated With Changes in Prefrontal Hemodynamics: a 3-armed Randomized Controlled Functional Near Infra-red Spectroscopy (fNIRS) Study
Brief Title: Neurophysiological Effects of Mind-body Exercise in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Yvonne Han, Associate Professor, Department of Rehabilitation Sciences, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20230213007
Record Dates: First submitted 2024-02-27; First posted 2024-03-29 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: mind-body practice; Qigong; Neurophysiology; Functional Near Infra-red Spectroscopy; fNIRS; Executive Function
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baduanjin Qigong(BDJ) (Experimental)
  Interventions: Behavioral: Baduanjin
- Aerobic exercise (Active Comparator)
  Interventions: Behavioral: Exercise
- Video viewing (Sham Comparator)
  Interventions: Behavioral: Video Viewing

INTERVENTIONS:
Behavioral: Baduanjin — The treatment group will individually perform single-session Baduanjin by following a video broadcasted the standardised BDJ protocol, which lasted for 12 minutes including 6 times of BDJ movements. Breathing rhythm is emphasised to be followed by participants.
  Other Names: Eight-Section Brocades Practice
  Arms: Baduanjin Qigong(BDJ)
Behavioral: Exercise — The active control group will individually perform 8-sets of aerobic exercise movement by following a video selected by registered physiotherapist.
  Arms: Aerobic exercise
Behavioral: Video Viewing — The control group will individually watch a 12-minute video with 6-minute introducing BDJ practice and 6 minute introducing aerobic exercise. This control group is used for controlling the effect of behavioural movement and brain activity generated by passive video viewing.
  Arms: Video viewing

SUMMARY:
There is some clinical evidence showing that Baduanjin (BDJ) practice, a type of mind-body based physical exercise, can improve executive function (EF). However, the neurophysiological changes associated with improved cognitive function remain elusive. Therefore, this study aims to carry out randomised controlled trial to explore how the single-session BDJ practice affect the function of prefrontal cortex(PFC) and also the EF of healthy adults, measure by fNIRS and verbal fluency test accordingly. A total of 60 healthy adults (based on power analysis 80% (β= 0.20) chance (α = 0.05, two-tailed)), aged 18 to 40 year old, without any physical, neurological, and neuropsychiatric disorder, classified as right-handed by Edinburgh Handedness Inventory, also with normal intelligence as verified by the Test of Nonverbal Intelligence will be recruited and randomly assigned to treatment(i.e. BDJ), active control(i.e, exercise), and passive control(i.e. video viewing) group. The investigator anticipate that this single-session BDJ practice will result in - (1) enhancing executive functioning , and (2) changes in functional brain activation pattern in PFC in adults. The result will give a spotlight to neurophysiological treatment effect of single-session Baduanjin on healthy adults, in developing intervention for improving executive functioning of adults.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed adults with normal intelligence (i.e. intelligence quotient ≥ 80), and without any physical, neuropsychiatric, and neurological disorders

Exclusion Criteria:

* Current positive history of head injury, seizure, stroke, other central nervous system diseases, other comorbid psychiatric illness, or reports of strong suicidal ideation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function as assessed by verbal fluency task (VFT) | 17 min after baseline
  Verbal fluency task (VFT). Executive functions are measured using the VFT. The experimental design of this task is adapted from previous fNIRS studies of verbal fluency where task blocks were interleaved with control blocks. Participants are required to generate exemplars of two semantic categories (i.e., animal and means of transportation) as many as possible, each for one minute, during the task blocks. This experimental task will begin with a 30-second phrase repetition period as a control, followed immediately by a 60-second task period (i.e, animal words), a 60-second control period, another 60-second task period (i.e., transportation words), and ended with another 60-second control period. The total measurement period is 270 seconds. The total number of correct and unique responses will be computed to reflect their fluency ability.
Hemodynamic changes as assessed by fNIRS | Baseline, during the 12-min intervention(immediate after baseline), immediate post-assessment(12 min after baseline)
  NIRSIT Lite is a portable, non-invasive neuroimaging procedure used to measure hemodynamic changes, in terms of oxyhemoglobin (HbO), deoxyhemoglobin (HbR) and total hemoglobin (HbT), associated with neuronal activities of the cerebral cortex in response to attending a task within the given period of time. Optical signals will be recorded on a two-wavelength (780 and 850 nm), continuous-wave optical imaging system (NIRSIT Lite; OBELAB Co., Seoul, South Korea). The 15 channels with a 30-mm source-detector separation which cover the entire PFC area will be used in this study. In accordance with the international 10-20 EEG system, the center of the bottom probe row will be placed at the reference point Fpz. Consequently, channel 1 to channel 7 represent the right PFC, and channel 9 to channel 15 the left PFC. In addition, NIRSIT has an embedded gyroscope that enables online removal of motion artifacts.

CONTACTS AND LOCATIONS:
Overall Officials: Hector Tsang, PhD, Study Chair — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong